CLINICAL TRIAL: NCT06704152
Title: A Phase 1/2a Multicenter Ascending Dose Study to Evaluate the Safety of HA-1 Minor Histocompatibility Antigen-Reactive TCR-Modified T Cells (BSB-1001) in Patients Undergoing HLA-Matched Allogenic Hematopoietic Stem Cell Transplant for AML, ALL or MDS
Brief Title: BSB-1001 in Patients Undergoing HLA-Matched Allogenic Hematopoietic Stem Cell Transplant for AML, ALL or MDS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BlueSphere Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BSB1001-CL-101
Record Dates: First submitted 2024-11-22; First posted 2024-11-25 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: AML, Adult Recurrent; ALL, Recurrent, Adult; MDS
Keywords: TCR, T-cell therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation Cohorts (Experimental): AML, ALL and MDS HLA-A*02:01 and HA-1-positive (H/H or H/R) patients with an identified HLA-matched, HA-1-negative (R/R) donor will be dosed in dose escalation cohorts
  Interventions: Drug: SOC + BSB-1001 Dose Escalation Cohort
- BSB-1001 Expansion Dose (Experimental): Once the maximum tolerated dose (MTD) or promising dose is reached additional AML HLA-A*02:01 and HA-1-positive (H/H or H/R) patients with an identified HLA-matched, HA-1-negative (R/R) donor will be enrolled in the expansion cohort.
  Interventions: Drug: SOC+BSB-1001 Expansion Dose

INTERVENTIONS:
Drug: SOC + BSB-1001 Dose Escalation Cohort — Patients will receive BSB-1001 a single intravenous (IV) infusion on day 0 following the infusion of the CD34-allo hematopoietic stem cell transplant (HCT).
  Arms: Dose Escalation Cohorts
Drug: SOC+BSB-1001 Expansion Dose — Patients will receive BSB-1001 a single intravenous (IV) infusion on day 0 following the infusion of the CD34-allo hematopoietic cell transplant (HCT).
  Arms: BSB-1001 Expansion Dose

SUMMARY:
The goal of this clinical trial is to test BSB-1001 which is a new type of cellular therapy to treat blood cancers (AML, ALL and MDS). It will evaluate the safety of BSB-1001 and also determine whether it works to prevent relapse of your cancer.

DETAILED DESCRIPTION:
This is a first-in-human, multicenter, open-label, dose-finding study for the evaluation of an HA-1 minor histocompatibility antigen (miHA)-reactive TCR-modified T cell product (BSB-1001) derived from an HLA-matched allogenic donor, in patients with AML, ALL or MDS undergoing an HLA-matched alloHSCT who are at a high risk for relapse post-HSCT. BSB-1001 targets the HLA-A*02:01-restricted HA-1 miHA.

Enrolled patients must be HLA-A*02:01 and HA-1-positive (H/H or H/R), with an identified HLA-matched, HA-1-negative (R/R) donor. Patients will undergo one of the following myeloablative conditioning regimens, according to standard institutional procedures, which include either fludarabine+thiotepa+total body irradiation, or busulfan+ melphalan+ fludarabine. After conditioning is completed, patients will receive the CD34-selected alloHSCT followed by BSB-1001 on day 0, without any prophylactic immunosuppression.

The study is an adaptive dose escalation design with 1 to 3 cohorts to evaluate single doses of BSB-1001. Three to six patients will be enrolled in each cohort and enrolled patients will be followed until completion of the study.

If the maximum tolerated dose (MTD) is reached or if a dose is deemed promising, the Sponsor may determine to either cease enrollment or open an expansion cohort at the desired dose level. The optional expansion part of the study is planned to include approximately 20 additional AML patients at the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ages 18 - 70 years inclusive, undergoing alloHCT.
2. Any of the following high-risk hematologic malignancies:

   1. AML diagnosed which has been treated with at least two lines of therapy* Refractory or relapsed (CR, CRh or CRi,), including myeloblasts up to 25% OR MRD positive OR persistent disease-defining cytogenetic abnormality OR MRD-negative, but with high-risk disease For patients in remission meeting criteria a, consolidation regimens would be considered another line of therapy of eligibility purposes
   2. ALL which has been with abnormal lymphoblasts ≥5% and up to 25% in bone marrow OR persistent disease-defining cytogenetic abnormality or MRD positive
   3. MDS after at least one line of therapy, which includes hypomethylating agent(s) and must be high or very high risk by Revised International Prognostic Scoring System (IPSS-R), monosomy, or complex karyotype or TP53 mutation.
   4. In the expansion phase AML patients diagnosed which has been treated with at least two lines of therapy, and refractory or relapsed (CR, CRh or CRi,), including myeloblasts up to 25% OR MRD positive OR persistent disease-defining cytogenetic abnormality OR MRD-negative, but with high- risk disease
3. HLA-A*02:01 AND HA-1 positive (either H/H or H/R).
4. Suitable for one of the approved conditioning regimens as defined in the protocol.
5. Patient must have an identified donor that is HA 1-negative with 10/10 matched related or unrelated donor

Exclusion Criteria:

1. Weight > 100 kg.
2. Prior history of allogeneic stem cell transplantation
3. Prior history of autologous stem cell transplantation within 1 year prior to the planned dosing of BSB-1001 (day 0)
4. Previous genetically engineered chimeric antigen receptor T Cell therapy (CAR-T), approved or investigational, within 2 years of screening, with the exception of patients with ALL previously treated with an autologous CAR-T product.
5. Treatment with other investigational agents within 5 half-lives of the planned dosing of BSB-1001 (day 0).
6. History of treatment with checkpoint inhibitor therapy within 3 months of transplantation.
7. Other malignancy with life expectancy < 1year.
8. Pregnant or lactating women.
9. Uncontrolled bacterial, viral, or fungal infections at time of enrollment.
10. Past or current viral infections as defined in the protocol.
11. CNS involvement refractory to intrathecal chemotherapy and/or standard cranial- spinal radiation. 12 Karnofsky Performance Score < 60%.

13. Inadequate organ function as defined in protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs), including SAEs, GVHD and dose-limiting toxicities | 365 days
  Incidence of TEAEs (per Common Terminology Criteria for Adverse Events [CTCAE])
Cellular kinetics of BSB-1001 in peripheral blood | 365 days
  Quantitation of BSB-1001 (copies per μL of genomic DNA)

SECONDARY OUTCOMES:
Number of patients with relapse | Through 365 days post HSCT
  Presence of malignant cells in marrow (>5%), peripheral blood (>1%), or extramedullary sites by histopathology after achievement of CR, CRh or CRi at any time after HSCT
Incidence of Grades II-IV acute GVHD | Through 100 days post HSCT
  Acute GVHD will be graded and assessed for response based on the MAGIC consortium scoring system
Incidence of Grades III-IV acute GVHD | Through 100 days post HSCT
  Acute GVHD will be graded and assessed for response based on the MAGIC consortium scoring system
Time to neutrophil engraftment | Through 365 days post HSCT
  Time to the first of 3 consecutive days of absolute neutrophil counts ≥ 500/µL
Time to platelet engraftment | Through 365 days post HSCT
  Time to ≥ 50,000/µL platelets for the first of 3 consecutive days without transfusion
Incidence of moderate to severe chronic GVHD | Through 365 days post HSCT
  Moderate-to-severe chronic GVHD graded according to NIH scale
Overall survival | Through 365 days
  Defined as the time from treatment to death due to any cause
GVHD-free, relapse-free survival (GFRS) | Through 365 days post HSCT
  Defined as time to any of the following events: 1) Grade III-IV aGVHD; 2) chronic GVHD requiring systemic immunosuppression; 3) primary malignancy relapse; or 4) death
GVHD-free survival (GFS) | Through 365 days post HSCT
  Defined as time to any of the following events: 1) GVHD event or 2) death from any cause
Incidence of systemic infections | Through 365 days post HSCT
  Defined as infections with a severity of Grades 3 to 5 (as graded by CTCAE v 5.0 or higher) which require treatment with systemic anti-infectives

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University at St Louis, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No